CLINICAL TRIAL: NCT01637012
Title: Prospective, Single-arm, Multicenter Study for Evaluation the Safety and Effectiveness of the ALEX Stent in a Real-world Setting of Percutaneous Coronary Interventions in Patients With Coronary Heart Disease. Study With Angiography and OCT Follow-up.
Brief Title: Prospective, Single-arm, Multicenter Study for Evaluation the Safety and Effectiveness of the ALEX Stent in a Real-world Setting of Percutaneous Coronary Interventions in Patients With Coronary Heart Disease
Acronym: ALEX OCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Balton Sp.zo.o. (Industry)
Collaborators: KCRI (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2.0, 2011-12-01
Record Dates: First submitted 2012-07-06; First posted 2012-07-10 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Stable Angina; Unstable Angina; Myocardial Infarction
Keywords: ALEX; coronary stent; cobalt-chromium; sirolimus; OCT
MeSH Terms: conditions — Angina, Stable; Angina, Unstable; Myocardial Infarction | interventions — Drug Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ALEX stent arm (Experimental): implantation of ALEX stent during index procedure
  Interventions: Procedure: Implantation

INTERVENTIONS:
Procedure: Implantation — index angioplasty with ALEX stent implatation
  Other Names: ALEX Stent

SUMMARY:
To evaluate the safety and effectiveness of the ALEX stent in a real-world setting of percutaneous coronary interventions in patients with coronary heart disease.

DETAILED DESCRIPTION:
Prospective, multicenter, non-randomized study designed to enroll up to 60 subjects to evaluate the safety and effectiveness of the cobalt-chromium sirolimus eluting coronary stent ALEX in a real-world setting of percutaneous coronary interventions in patients with coronary heart disease.

ELIGIBILITY:
Inclusion Criteria:

Clinical Inclusion Criteria:

* > 18 years of age
* Patient must provide written informed consent prior to procedure using a form that is approved by the local Ethics Committee
* clinical diagnosis of Stable Angina, Unstable Angina or Myocardial Infarction without ST elevation (NSTEMI) or Myocardial Infarction with ST elevation provided the expiry of 72 hours of the onset of symptoms and stable clinical and hemodynamical condition the Patient with patent postinfarcion artery (TIMI 3) and indications for PCI and next stage of revascularization in the other vessels
* earlier effective supply of others lesions in others vessels in case of multivessels disease
* female of childbearing potential must have a negative pregnancy test within 7 days prior to enrolment and utilize reliable birth control for 12 months after enrolment

Angiographic Inclusion Criteria

* target lesion stentosis must be > 70% (visual estimate)
* Patient eligible for PCI treatment with the ALEX stent system (vessel diameter in range of 2.5 to 4.0 mm and length of lesion that allows to cover a single stent with maximum length of 30 mm in visual evaluation)

Exclusion Criteria:

Clinical Exclusion Criteria

* anticipated inablility of the patient to comply with 12 months of antiplatelet treatment (e. g. elective non-cardiac surgery following stenting, drug intolerance etc.)
* acute or chronic renal failure (serum creatinine > 2 mg%, GFR < 60 ml/min/1.73m2)
* left ventricular ejection fraction (LVEF) < 40%
* cardiogenic shock
* short life expectancy (< 1 year)
* any significant medical condition which in the investigator's opinion may interference with the Patient's optimal participation in the study
* current participation in another drug or device clinical trail in which there no be reached the primary endpoint or which clinically interferences with trail's enpoints

Angiographic Exclusion Criteria

* chronic total occlusion
* calcified lesion which cannot be successfully dilated
* location of lesions in the winding vessels where there is no possibility of OCT imaging
* target stenosis located in venous or arterial bridge
* unprotected left main coronary disease with > 50% stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Assessment of stent strut coverage and parameters of restenosis | at 12 months follow-up
  Assessment of stent strut coverage and parameters of restenosis in coronary angiography (QCA - Late Lumen Loss) and in OCT (percent of neointimal volume) 12 months follow-up after the baseline procedure in group of first 20 patients
Assessment of stent strut coverage and parameters of restenosis | at 6 months follow-up
  Assessment of stent strut coverage and parameters of restenosis in coronary angiography (QCA - Late Lumen Loss) and in OCT (percent of neointimal volume) 6 months follow-up after the baseline procedure in group of second 20 patients
Assessment of stent strut coverage and parameters of restenosis | at 3 months follow-up
  Assessment of stent strut coverage and parameters of restenosis in coronary angiography (QCA - Late Lumen Loss) and in OCT (percent of neointimal volume) at 3 months follow-up after the baseline procedure in group of third 20 patients

SECONDARY OUTCOMES:
Procedural success | during index hospitalization
  Procedural success during baseline PCI assessed in coronary angiography (QCA)
Occurrence of stent thrombosis | at 30 days follow-up
  Occurrence of stent thrombosis at 30 days follow-up
Occurrence of stent thrombosis | at 12 months follow-up
  Occurrence of stent thrombosis at 12 months follow-up
Incidence of Major Adverse Cardiac Events | at 30 days follow-up
  Incidence of Major Adverse Cardiac Events (MACEs) at 30 days follow-up defined as death, myocardial infarction target lesion re-PTCA or target lesion bypass graft
Incidence of Major Adverse Cardiac Events | at 12 months follow-up
  Incidence of Major Adverse Cardiac Events (MACEs) at 12 months follow-up defined as death, myocardial infarction target lesion re-PTCA or target lesion bypass graft

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Legutko, MD, PhD, Principal Investigator — Szpital Uniwersytecki w Krakowie, ul. Kopernika 17, Krakow 31-501, Poland; Dariusz Dudek, Prof., Study Chair — Szpital Uniwersytecki w Krakowie, ul. Kopernika 17, Krakow 31-501, Poland
Locations (5):
- Poland (5):
  - Carint Scanmed Szpital Sw. Rafala, Krakow, Bochenka 12
  - Szpital Uniwersytecki w Krakowie, Samodzielna Pracownia Zakladu Hemodynamiki i Angiografii, Krakow, Kopernika 17
  - Polsko-Amerykanskie Kliniki Serca I Oddzial Kardiologiczno-Angiologiczny, Ustroń, Sanatoryjna 7
  - Polsko-Amerykanskie Kliniki Serca III Oddzial Kardiologii Inwazyjnej, Angiologii i Elektrokardiologii, Dąbrowa Górnicza, Szpitalna 13
  - Centralny Szpital Kliniczny MSWiA w Warszawie Klinika Kardiologii Inwazyjnej, Warsaw, Woloska 137

REFERENCES:
- See also: Sponsor — http://www.balton.pl/